CLINICAL TRIAL: NCT00399646
Title: Gemini Angioplasty and Arterial Measurement Evaluation (GAAME) An Evaluation of the Metricath Gemini System, a Percutaneous Interventional Device Intended to Make Arterial Lumen Measurements and Perform Percutaneous Transluminal Angioplasty Dilations.
Brief Title: Evaluation of the Metricath Gemini System, a Device Intended to Make Arterial Measurements and Perform Angioplasty Dilations.
Acronym: GAAME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Fabio De Pasquale, Regulatory Afairs Director, Neovasc, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: revJ060707
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2009-05-13 (Estimated); Status verified 2009-05

CONDITIONS: Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Metricath Gemini System

SUMMARY:
The purpose of the Metricath Gemini System is to pre-dilate the target treatment area, take arterial lumen measurements in a native section of artery or within the deployed stent and perform further dilation of the deployed stent if required. In this manner, the Metricath Gemini System can assist the Interventionalist by providing arterial measurements prior to stenting, performing pre-stenting angioplasty, taking within stent measurements to help determine if the stent is fully deployed, and by performing post-stenting dilations to further dilate the stent if required.

DETAILED DESCRIPTION:
Several recent clinical studies have suggested that proper vascular stent deployment directly affects clinical outcome, and the rate of re-stenosis. These studies suggest that angiography alone is not sufficient to ensure proper vascular stent deployment, and that re-stenosis rates will decline if proper stent apposition has occurred. The importance of proper stent sizing and apposition is further emphasised with the increasing use of drug eluting stents, the drug effects of which are only realized upon contact with the arterial wall.

Angiometrx Inc. developed the Metricath Arterial Measurement System in response to the need for increased stent sizing and deployment. The Metricath System measures the diameter and cross sectional area of arteries using an intravascular balloon catheter attached to a computerized console. Considering the ease and rapidity of obtaining Metricath results, this technique may form an alternative to evaluate vessel area and stent expansion.

The Metricath System was 510(k) cleared in the U.S. in June, 2003, and received European and Canadian market approvals in 2004.

Angiometrx Inc. has now developed the next generation of Metricath System, which incorporates a second balloon on the catheter, intended for angioplasty purposes. The Metricath Gemini System is comprised of a dual balloon catheter which is attached to the same Metricath computerized console as the Metricath System. As with the Metricath System, the Metricath Console operates the inflation and deflation of the Gemini measurement balloon and provides arterial cross-sectional area and diameter. The Metricath Gemini angioplasty balloon is controlled separately in the traditional manner using a hand-held inflation device, attached to a port in the hub of the catheter.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom coronary artery angiography is indicated and angioplasty and stenting is being considered.
* Single vessel disease of an artery with a lesion assessable to standard coronary guidewires and are scheduled or indicated for percutaneous coronary intervention.
* A maximum of one lesion requiring treatment (angioplasty +/- stenting) to an intended arterial diameter of 2.5 mm - 4.0 mm.
* Target stent length of 15 mm - 32 mm, where a single stent can adequately cover the lesion.
* Stenotic de novo lesions in native coronary arteries.

Exclusion Criteria:

* Women who are pregnant.
* Participation in a study involving investigational drugs or devices during the last six months.
* Patients with previous stenting in the target vessel area.
* Patients who experienced a myocardial infarction, Braunwald Class C, and very unstable Braunwald Class B3 within 6 weeks prior to the procedure or have unstable angina pectoris.
* Patients who are experiencing TIA's or minor or major strokes within six months prior to procedure.
* Contraindicated for antiplatelet and/or anticoagulation medications.
* Symptoms of cardiogenic shock.
* Patients who underwent a staged procedure 30 days prior to enrolment and/or were scheduled to have a staged procedure 14 days after treatment.
* Significant liver or kidney disease or malignancy.
* Patients scheduled for any other surgery or other procedure within 30 days.
* Severe peripheral vascular disease preventing femoral access.
* Left ventricle ejection fraction of < 35%.
* Total occlusion of target vessel.
* A blood pressure in excess of 180 mmHg at the time of the angiography.
* Visible thrombus, filling defect, or ulceration in the target artery.
* Severely calcified lesions which suggest that balloon pre-dilatation will not achieve adequate luminal diameter to allow successful stent delivery and deployment.
* The target lesion is beyond a left main artery stenosis > 50%.
* Contraindicated for CABG.
* Coronary spasm in the absence of a significant stenosis.
* Requiring treatment of more than two lesions.
* Requiring treatment with atherectomy.
* Lesions in surgical conduits - saphenous vein grafts, internal mammary arteries, or radial arteries.
* Unprotected left main coronary artery.
* Diffuse disease.
* Excessive tortuosity of proximal segment.
* Extremely angulated segments > 90°.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2005-11; Primary Completion 2007-11 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To observe the safety of the device, as determined by freedom from MACE (major adverse cardiac events) within 30 days post-procedure. | 30 days
To observe the success of the device as determined by residual diameter stenosis | 30 days
To evaluate the inflation of dilation balloon to desired pressure | immediate

SECONDARY OUTCOMES:
To evaluate the successful delivery of catheter to target area | immediate
To evaluate the performance of the device to measure arterial size | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Willem van der Giessen, MD, Principal Investigator — Department of Cardiology, Thoraxcenter, Erasmus Medical Center, The Netherlands; Evelyn Regar, MD, Principal Investigator — Department of Cardiology, Thoraxcenter, Erasmus Medical Center, The Netherlands; David Kandzari, MD, Principal Investigator — Division of Cardiology and Duke Clinical Research Institute, Duke University Medical Center, USA
Locations (16):
- United States (10):
  - UC Irvine Medical Center, Orange, California
  - Mercy Heart Institute, Sacramento, California
  - Pasco Cardiology Center, Hudson, Florida
  - Baptist Miami Hospital, Miami, Florida
  - Florida Cardiovascular Institute, Tampa, Florida
  - Sinai Hospital, Baltimore, Maryland
  - Columbia Presbyterian Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Tyler Cardiovascular Consultants, Tyler, Texas
- Canada (2):
  - Vancouver Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
- Netherlands (4):
  - Amphia Hospital, Breda, The Netherlands
  - Leiden University Medical Center, Leiden, The Netherlands
  - Medisch Centrum Rijmond Zuid, Rotterdam, The Netherlands
  - University Medical Center Rotterdam, Rotterdam, The Netherlands

REFERENCES:
- [Background] de Jaegere P, Mudra H, Figulla H, Almagor Y, Doucet S, Penn I, Colombo A, Hamm C, Bartorelli A, Rothman M, Nobuyoshi M, Yamaguchi T, Voudris V, DiMario C, Makovski S, Hausmann D, Rowe S, Rabinovich S, Sunamura M, van Es GA. Intravascular ultrasound-guided optimized stent deployment. Immediate and 6 months clinical and angiographic results from the Multicenter Ultrasound Stenting in Coronaries Study (MUSIC Study). Eur Heart J. 1998 Aug;19(8):1214-23. doi: 10.1053/euhj.1998.1012. PMID 9740343
- [Background] Fitzgerald PJ, Oshima A, Hayase M, Metz JA, Bailey SR, Baim DS, Cleman MW, Deutsch E, Diver DJ, Leon MB, Moses JW, Oesterle SN, Overlie PA, Pepine CJ, Safian RD, Shani J, Simonton CA, Smalling RW, Teirstein PS, Zidar JP, Yeung AC, Kuntz RE, Yock PG. Final results of the Can Routine Ultrasound Influence Stent Expansion (CRUISE) study. Circulation. 2000 Aug 1;102(5):523-30. doi: 10.1161/01.cir.102.5.523. PMID 10920064
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Background] Cannon CP, Battler A, Brindis RG, Cox JL, Ellis SG, Every NR, Flaherty JT, Harrington RA, Krumholz HM, Simoons ML, Van De Werf FJ, Weintraub WS, Mitchell KR, Morrisson SL, Brindis RG, Anderson HV, Cannom DS, Chitwood WR, Cigarroa JE, Collins-Nakai RL, Ellis SG, Gibbons RJ, Grover FL, Heidenreich PA, Khandheria BK, Knoebel SB, Krumholz HL, Malenka DJ, Mark DB, Mckay CR, Passamani ER, Radford MJ, Riner RN, Schwartz JB, Shaw RE, Shemin RJ, Van Fossen DB, Verrier ED, Watkins MW, Phoubandith DR, Furnelli T. American College of Cardiology key data elements and definitions for measuring the clinical management and outcomes of patients with acute coronary syndromes. A report of the American College of Cardiology Task Force on Clinical Data Standards (Acute Coronary Syndromes Writing Committee). J Am Coll Cardiol. 2001 Dec;38(7):2114-30. doi: 10.1016/s0735-1097(01)01702-8. No abstract available. PMID 11738323
- [Background] Smith SC Jr, Dove JT, Jacobs AK, Kennedy JW, Kereiakes D, Kern MJ, Kuntz RE, Popma JJ, Schaff HV, Williams DO, Gibbons RJ, Alpert JP, Eagle KA, Faxon DP, Fuster V, Gardner TJ, Gregoratos G, Russell RO, Smith SC Jr; American College of Cardiology/American Heart Association task force on practice guidelines (Committee to revise the 1993 guidelines for percutaneous transluminal coronary angioplasty); Society for Cardiac Angiography and Interventions. ACC/AHA guidelines for percutaneous coronary intervention (revision of the 1993 PTCA guidelines)-executive summary: a report of the American College of Cardiology/American Heart Association task force on practice guidelines (Committee to revise the 1993 guidelines for percutaneous transluminal coronary angioplasty) endorsed by the Society for Cardiac Angiography and Interventions. Circulation. 2001 Jun 19;103(24):3019-41. doi: 10.1161/01.cir.103.24.3019. No abstract available. PMID 11413094
- [Background] van der Giessen WJ, Regar E, McFadden E, McDougall I, Serruys PW. Assessment of stent dimensions with a novel intracoronary balloon-based system: comparative study versus intravascular ultrasound and quantitative coronary angiography. The CAMUS - Coronary Angioplasty Metricath vs. UltraSound Trial. EuroIntervention. 2005 Aug;1(2):244-51. PMID 19758910